CLINICAL TRIAL: NCT00006273
Title: Study of Total Energy Expenditure in Infants and Children With Moderate to Severe Cystic Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Indiana University School of Medicine (Other)
Other Study IDs: NCRR-M01RR00750-9040; IU-9509-20
Record Dates: First submitted 2000-09-11; First posted 2000-09-12 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Cystic Fibrosis
Keywords: cardiovascular and respiratory diseases; cystic fibrosis; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
OBJECTIVES: I. Compare the resting energy expenditure using respiratory calorimetry in infants and children with moderate to severe cystic fibrosis versus age matched healthy controls.

II. Determine the total energy expenditure and energy spent on physical activity using the doubly labeled water method in these patient populations.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients and healthy controls receive an oral dose of doubly labeled water following initial urine collection on day 1. Patients undergo additional urine collection at 4-6 hours following doubly labeled water consumption and then daily for 7 days.

Additionally, at the beginning of the study, patients and healthy controls undergo respiratory calorimetry over approximately 45 minutes at rest, starting approximately 2-3 hours after the last meal consumption and last use of aerosol bronchodilators (if required).

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of cystic fibrosis (CF) by two positive sweat tests No exacerbations of present condition within past 2 months FEV1 less than 50% of predicted No other uncorrected lung disease No requirement for supplemental oxygen

OR

* Healthy (control group) Age matched to CF patients No preexisting lung disease Clinically well No hospitalizations within past 6 months

--Prior/Concurrent Therapy--

* Concurrent pancreatic enzyme supplementation for CF required Clinically stable on current medications (CF patients)

--Patient Characteristics--

* Age: Birth to 12 months 6 to 10 years
* Cardiovascular: No major cardiovascular problems (CF patients) No preexisting heart disease (control group)
* Pulmonary: See Disease Characteristics
* Other: No chromosomal abnormalities (CF patients) No acute infection (CF patients) No diabetes mellitus (both groups)

Ages: 0 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60
Dates: Start 1996-06

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A. Leitch, Study Chair — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States